CLINICAL TRIAL: NCT06458270
Title: Perceived Effectiveness of Salt Warning Labels on a UK Restaurant Menu: a Real-world Pilot Experiment
Brief Title: Salt Warning Label Restaurant Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Eric Robinson, Professor Eric Robinson, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: rfj78drdsu52lsbw3kztnbpne8xdao
Record Dates: First submitted 2024-06-03; First posted 2024-06-13 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Food Selection
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Label group (Experimental): Participants will receive a manipulated restaurant menu featuring salt warning labels next to menu items that are high in salt.
  Interventions: Behavioral: Salt warning label
- Control group (no label) (No Intervention): Participants will receive a standard restaurant menu (no labels).

INTERVENTIONS:
Behavioral: Salt warning label — A salt warning label will feature on the restaurant menu next to menu items that are high in salt (>3g, more than 50% of guideline daily amount [GDA] in the UK).
  Arms: Label group

SUMMARY:
This between-subjects randomised controlled trial aims to test the effect of a menu featuring salt warning labels on perceived message effectiveness relative to a menu with no labels in a real-world restaurant environment. The study will also act as a pilot experiment for examining the impact of the salt warning label on food choice and subsequent salt intake in real-world conditions.

Primary objectives:

* To measure the PME of a menu featuring salt warning labels relative to a menu with no labels
* To measure label awareness, perceived knowledge gain, and perceived influence of the label on food choice

Secondary objectives:

* To identify whether there is an effect of the salt warning label on:

  * Food choice (label/no label)
  * Total salt selected
  * Total salt intake
* To examine support for the introduction of a salt warning label policy in the UK

ELIGIBILITY:
Inclusion Criteria:

* Are a UK resident
* Are aged 18 years and above
* Are fluent in English
* Eat an out-of-home meal at least once a month on average
* Have no dietary allergies
* Are not vegan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2024-09-14 (Actual); Study Completion 2024-09-14 (Actual)

PRIMARY OUTCOMES:
Perceived message effectiveness (PME) | Post - meal assessment (within 10 minutes)
  Participants will answer 3 PME questions using a Likert scale ranging from 1 - 5 anchored by "not at all" and "a great deal": Prompt: "Think back to the menu that you ordered from…" "The menu made me concerned about the health effects of consuming items high in salt", "The menu made consuming items high in salt seem unpleasant", "The menu discouraged me from wanting to consume items high in salt". The mean response to the three items will be calculated.
Label awareness | Post - meal assessment (within 10 minutes)
  "Did you notice any warning labels next to any of the menu items when making your meal selection?" (yes/no).
  If [yes], "What did the label tell you about?" Response options: Healthy items, Organic, Calcium, Sustainable, Added sugars, Vegetarian, Unhealthy items, Salt, Fibre, Gluten Free, None of these, Not sure.
  If [yes], "Please describe what the label said" (open text response). Responses that mention high in salt or similar will be coded as aware.
Salt awareness | Post - meal assessment (within 10 minutes)
  "Did you think about the salt content of the meals when making your selection?" (yes/no)
Perceived knowledge gain | Post - meal assessment (within 10 minutes)
  For this question, both conditions will be shown an image of the labelled menu. "Did you learn something new from the salt labels on the menu?" (yes/no).
Perceived influence | Post - meal assessment (within 10 minutes)
  For this question, both conditions will be shown an image of the labelled menu, and some question phrasing is slightly altered.
  "Did the salt label influence which food you ordered from the menu" (yes/no). "If [yes], how did the salt label influence your choice?" Response options: I avoided choosing a meal high in salt; I chose a meal high in salt; Other (free text response) Control: "Would the salt label have influenced what food you ordered from the menu?" (yes/no) If [yes], how would the salt label have influenced your choice? Response options: I would have avoided choosing a meal high in salt; I would have chosen a meal high in salt; Other (free text response)
Policy support | Post - meal assessment (within 10 minutes)
  For this question, the both conditions will be shown an image of the labelled menu.
  If the UK Government introduced policy requiring restaurant menu items high in salt to feature these labels, how would you feel?" Likert scale ranging from 1 - 5 anchored by "strongly oppose" and "strongly support".

SECONDARY OUTCOMES:
Total salt purchased | Post - meal assessment (within 10 minutes)
  Determined based on the total order of the participant, including food and drink. Prior to study commencement, all menu items will be sent for nutritional analysis to determine salt content/100g. Menu items will be weighed before being sent for analysis using kitchen scales (Vitafit VT706), so that specific salt content per serving can be calculated.
Labelled item selected | Post - meal assessment (within 10 minutes)
  Determined based on whether the food item selected featured a high in salt warning label (yes = 1, no = 0).
Total salt consumed | Post - meal assessment (within 10 minutes)
  Salt consumption will be determined from the order that the researcher takes and an estimation of the proportion of the meal that was consumed. The researcher will take a photograph before and after consumption and will estimate the percentage consumed component(s) of the meal, taking into account whether participants leave a proportion of all meal components or specific components (e.g., low salt or high salt components). Participants will also be asked whether they shared any of their meal with someone else. A random 10% selection of percentage estimates will be performed by a second researcher to measure reliability. Food consumption will then be calculated by subtracting an estimation of the proportion of the meal that was consumed (taking into account if any has been shared) from the food purchase.
Later salt intake | Follow-up assessment (next morning, 8AM, to be completed within 24 hours)
  Participants will receive a link to a dietary recall questionnaire (Intake24, https://intake24.co.uk/) via email on the same day after taking part in the study, which they will be prompted to complete before bed. They will be asked to provide as much detail as possible on what they had for dinner, snacks, and drinks after the restaurant visit. Based on this information and salt values calculated by Intake24, the total salt consumed by the participants for the rest of the day after the visit will be estimated.
Other macronutrient intake | Post - meal assessment (within 10 minutes)
  Total kcal, sugar, and saturated fat intake [i.e., other nutrients that are not the main warning focus] will be calculated based on the nutritional content of the order of the participant.

OTHER OUTCOMES:
Food choice motives | Post - meal assessment (within 10 minutes)
  The "health" subsection of the Food Choice Questionnaire will be used to measure the extent to which health motives may influence participants' food choices. The subsection consists of 6 items, e.g. "It is important to me that the food I eat on a typical day….is nutritious" answered on a 4-point Likert scale ranging from "Not at all important" to "Very important". The mean response for the six items will be calculated.
Aim guessing | Post - meal assessment (within 10 minutes)
  Participants are told that the study is about dining habits in restaurants. At the start of the post-meal assessments, participants will be asked what they think the aims of the study were (free text response). Any participant that guesses the study aims to be investigating the influence of food warning labels on food choice will be coded as being aware of study aims. One researcher will code awareness of aims (R.E.) and a second researcher will independently verify the coding.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liverpool, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The anonymised dataset has been uploaded to the Open Science Framework (OSF) - https://osf.io/whzc8/?view_only=e97eb9ff6812457081d6d693e27bf1bd
Supporting Information: Study Protocol, SAP, ICF, Analytic Code

REFERENCES:
- [Derived] Evans R, Brealey J, Clarke N, Falbe J, Finlay A, Jones A, Thorp P, Witham B, Witkam R, Robinson E. Salt warning labels in the out-of-home food sector: online and real-world randomised controlled trials in the UK. Lancet Public Health. 2025 Aug;10(8):e656-e667. doi: 10.1016/S2468-2667(25)00143-4. PMID 40738552

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT06458270/Prot_SAP_ICF_000.pdf